CLINICAL TRIAL: NCT06550856
Title: SUTURE-CLOSURE OMENTOPEXY VERSUS OMENTOPEXY ALONE IN REPAIR OF PERFORATED PEPTIC ULCER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Adel Ashraf Abdrabou, Resident in the Department of General Surgery, oncological and Laparoscopic Surgery Sohag University Hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-07-07MS
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Perforated Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUTURE-CLOSURE OMENTOPEXY IN REPAIR OF PERFORATED PEPTIC ULCER (Active Comparator): Group (A ) includes modification of the Graham's patch will be used in this group, where suitable sutures are passed between the edges of perforation and tied to close the perforation. A pedicle of omentum based on right omental artery is brought between these sutures, and these sutures are tied again with pedicle of omentum between knots over the perforation (thus the omentum remains sandwiched between the two levels of secured knots).
  Interventions: Procedure: SUTURE-CLOSURE OMENTOPEXY IN REPAIR OF PERFORATED PEPTIC ULCER
- OMENTOPEXY ALONE IN REPAIR OF PERFORATED PEPTIC ULCER (Active Comparator): Group (B) includes Grahm's technique of omentopexy will be performed by closing the perforation by placing interrupted full thickness suitable sutures along the margins of the ulcer with a patch of pedicled omentum laid over these sutures, which are then tied (without any attempt for primary closure of the perforation before placing the omentum as a plug).
  Interventions: Procedure: OMENTOPEXY ALONE IN REPAIR OF PERFORATED PEPTIC ULCER

INTERVENTIONS:
Procedure: SUTURE-CLOSURE OMENTOPEXY IN REPAIR OF PERFORATED PEPTIC ULCER — Patients presented with perforated peptic ulcer will be repaired using full thickness suture closure using 3/0 vicryl suture then omental patch laied over the sutures.
  Arms: SUTURE-CLOSURE OMENTOPEXY IN REPAIR OF PERFORATED PEPTIC ULCER
Procedure: OMENTOPEXY ALONE IN REPAIR OF PERFORATED PEPTIC ULCER — Patients presented with perforated peptic ulcer will be repaired by using omental patch without any attempt for primary closure of perforation.
  Arms: OMENTOPEXY ALONE IN REPAIR OF PERFORATED PEPTIC ULCER

SUMMARY:
The present study will be conducted to assess whether there is a direct benefit associated with modified-Graham's omentopexy (MGO), above and beyond the benefit associated with Graham's omentopexy (GO) in the treatment of perforated duodenal ulcers. We attempted to answer the question whether primary closure of the perforation in MGO will affect the outcome of surgery. Complication rates will be compared for the two alternative surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

- All adult patients of both sexes with a clinical diagnosis of perforated peptic ulcer (gastric or duodenal) that are fit to undergo surgery.

Exclusion Criteria:

- 1. Patients with associated bleeding ulcer (additional steps are needed to control bleeding).

2. Patients with associated pathology other than perforated peptic ulcer that needs surgical intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Early postoperative follow up for repair of perforated peptic ulcer | Three days after the operation
  resumption of oral intake

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Berne TV, Donovan AJ. Nonoperative treatment of perforated duodenal ulcer. Arch Surg. 1989 Jul;124(7):830-2. doi: 10.1001/archsurg.1989.01410070084017. PMID 2742484
- [Background] Boey J, Choi SK, Poon A, Alagaratnam TT. Risk stratification in perforated duodenal ulcers. A prospective validation of predictive factors. Ann Surg. 1987 Jan;205(1):22-6. doi: 10.1097/00000658-198701000-00005. PMID 3800459
- [Background] Chung KT, Shelat VG. Perforated peptic ulcer - an update. World J Gastrointest Surg. 2017 Jan 27;9(1):1-12. doi: 10.4240/wjgs.v9.i1.1. PMID 28138363